CLINICAL TRIAL: NCT05662085
Title: Progression Rate of Pseudoxanthoma Elasticum-associated Choroidal and Retinal Degeneration
Acronym: PROPXE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: PROPXE
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Pseudoxanthoma Elasticum
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — According to clinical practice.

SUMMARY:
This study aims to systematically assess the retest reliability and ability to detect a change of new visual function tests and ophthalmological imaging methods for observing the natural course of pseudoxanthoma elasticum (PXE).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Pseudoxanthoma elasticum according to the Plomp criteria or adult patients with a PXE-mimicking phenotype (angioid streaks and peau d'orange [e.g., ENPP1 or GGCX-associated disease])
* Best-corrected visual acuity (BCVA): ≤1.0 LogMAR

Exclusion Criteria:

* Inability to give informed consent
* Claustrophobia
* Prior surgery (other than anti-VEGF injections, cataract surgery, YAG laser capsulotomy, or laser retinopexy) that - according to the investigator's judgment - may affect visual function assessments (e.g., retinal detachment surgery, glaucoma filtration surgery, or a history of a corneal transplant in the study-eye)
* Concurrent ophthalmic conditions in the study eye that (according to the investigator's judgment) may contribute to loss of vision, such as clinically significant opacification of the ocular media (corneal dystrophies, cataract), other retinal diseases, or disease of the optic nerve head and visual pathway (including amblyopia)
* Major surgery planned or other events that (according to the investigator's judgment) could hinder follow-up examinations (e.g., knee replacement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include subjects with PXE and PXE-mimicking ocular phenotypes.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in the rate of rod-mediated dark-adaptation at the leading disease front (i.e., change in the rod-intercept time [RIT in min] per year) | Two years from Baseline

SECONDARY OUTCOMES:
Change in Bruch's membrane reflectivity | Two years from Baseline
Change in choriocapillaris loss | Two years from Baseline
Change in steady-state rod and cone sensitivity | Two years from Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Pfau, MD, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hess K, Gliem M, Charbel Issa P, Birtel J, Muller PL, von der Emde L, Herrmann P, Holz FG, Pfau M. Mesopic and Scotopic Light Sensitivity and Its Microstructural Correlates in Pseudoxanthoma Elasticum. JAMA Ophthalmol. 2020 Dec 1;138(12):1272-1279. doi: 10.1001/jamaophthalmol.2020.4335. PMID 33090206
- [Background] Hess K, Gliem M, Birtel J, Muller P, Hendig D, Andrews C, Murray IJ, Holz FG, Charbel Issa P. IMPAIRED DARK ADAPTATION ASSOCIATED WITH A DISEASED BRUCH MEMBRANE IN PSEUDOXANTHOMA ELASTICUM. Retina. 2020 Oct;40(10):1988-1995. doi: 10.1097/IAE.0000000000002689. PMID 31834130
- [Background] Pfau K, Lengyel I, Ossewaarde-van Norel J, van Leeuwen R, Risseeuw S, Leftheriotis G, Scholl HPN, Feltgen N, Holz FG, Pfau M. Pseudoxanthoma elasticum - Genetics, pathophysiology, and clinical presentation. Prog Retin Eye Res. 2024 Sep;102:101274. doi: 10.1016/j.preteyeres.2024.101274. Epub 2024 May 28. PMID 38815804
- [Result] Pfau K, Ansari G, Michels S, Dysli C, Liakopoulos S, Burghaus-Zhang J, Al-Sheikh M, Garweg JG, Quinodoz M, Kaminska K, Cancellieri F, Rivolta C, Terry SF, Feltgen N, Pfau M. Topography of Slowed Dark Adaptation in Pseudoxanthoma Elasticum: PROPXE Study Report 1. Invest Ophthalmol Vis Sci. 2025 Feb 3;66(2):17. doi: 10.1167/iovs.66.2.17. PMID 39913163
- [Derived] Giger JAW, Ansari G, Terry SF, Charbel Issa P, Pfau K, Pfau M; PROPXE Study Group. Measurement Reliability and Functional Validity of Bruch's Membrane Calcification in Pseudoxanthoma Elasticum: PROPXE Study Report 2. Invest Ophthalmol Vis Sci. 2025 Nov 3;66(14):29. doi: 10.1167/iovs.66.14.29. PMID 41230901